CLINICAL TRIAL: NCT03910517
Title: Musculoskeletal Pain Among E-sport Athletes
Status: Completed | Type: Observational
Sponsor: University College of Northern Denmark (Other)
Responsible Party: Principal Investigator, Christian Lund Straszek, Assistant lecturer, University College of Northern Denmark
Other Study IDs: Project E-sport
Record Dates: First submitted 2019-03-26; First posted 2019-04-10 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-05

CONDITIONS: Musculoskeletal Pain
Keywords: Musculoskeletal Pain; Sleep; Training load; E-sport; Physical activity
MeSH Terms: conditions — Musculoskeletal Pain; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- E-sport athletes: People aged 15-35 who engage in structured E-sport (e.g. community-based, pro team or educational setting).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Background:

Musculoskeletal (MSK) pain and injuries are common in endurance sports where athletes are required to perform at high intensity for long periods of time. In the short term, MSK pain may significantly impair the athletes' performance, which can lead to unwanted time-off from practice and competitive tournaments. Previous studies found an association between training load, MSK pain and performance. These results indicate that an athlete may experience MSK pain or get injured from both too low and to high training loads.

Electronic sports (E-sports), also known as competitive gaming, is defined by Hamari and Sjöblom as "a form of sports where the primary aspects of the sport is facilitated by electronic systems; the input of players and teams as well as the output of the E-sports system are mediated by human-computer interference".

There are only few data on MSK pain in E-sports, however a small study with 65 participants found that 41% suffered from back or neck pain and more than 1 in 3 had pain related to the wrist. E-sports athletes have to perform for an extended period of time, similar to athletes from traditional endurance sport. As such, MSK pain in E-sports may be associated with training load like it is seen in other sports. Therefore, MSK pain in E-sports could be an unrecognised issue. To provide health professionals with and optimal starting point for managing these issues, there is a need for well-conducted studies on the prevalence of MSK pain among E-sports athletes. In addition, it is highly relevant to investigate if training loads related to E-sports and physical activity levels are different among athletes with MSK pain compared to athletes without MSK pain.

Aims:

The aims of this questionnaire-based cross-sectional study are to; I) investigate the prevalence of MSK pain in E-sports athletes, II) assess if training loads among athletes with MSK pain are different from athletes without MSK pain, III) investigate if physical activity levels among athletes with MSK pain are different from athletes without MSK pain and IIII) descriptively present data on participant characteristics, sleep patterns, physical activity levels and utilization of health professionals and pain medication in the study population.

DETAILED DESCRIPTION:
Data analysis:

The prevalence of MSK pain within the study population will be presented in absolute numbers and as percentage values. To investigate if E-sport related training loads differ among athletes with and without MSK pain we will use total E-sport related training load (N hours spend on structured E-sport + N hours spend on unstructured E-sport). An independent sample t-test will be applied for this comparison if data are normally distributed. To assess if physical activity levels are different among athletes with and without MSK pain we will use the responses from the IPAQ short form. For this comparison we will use an independent sample t-test or the Wilcoxon rank-sum test. Participant characteristics, distribution and number of MSK pain sites, utilization of health professionals and pain medicine, physical activity levels, training loads and sleep patterns will be presented descriptively. The data will be presented with means, standard deviations and 95% confidence intervals. Non-parametric data will be presented with absolute numbers and as percentage values, medians and range.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-35
* Engaged in E-sport at an educational institution, a community-based team or a pro-team.
* Participating in E-sport through a computer-based game.

Exclusion Criteria:

* Not providing written informed consent prior to enrolment.

Ages: 15 Years to 35 Years | Sex: All
Age Groups: Child, Adult
Study Population: People aged 15-35 who engage in E-sport at an educational institution, a community-based team or a pro-team in Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Prevalence of pain in the body during the previous week. | Baseline - at time of inclusion
  Participants are asked if they have experienced any pain in their body during the previous week (yes/no).

SECONDARY OUTCOMES:
Primary pain site: questionnaire | Baseline - at time of inclusion
  Participants are asked where in the body they experience their primary pain complaint (list: head, chest, stomach, back, neck, shoulder, upper arm, elbow, forearm, wrist, hand/fingers, hip/groin, thigh, knee, shinbone, ankle, and foot/toes).
Other pain sites: questionnaire | Baseline - at time of inclusion
  Participants are asked if they experience pain at additional sites (List: head, chest, stomach, back, neck. Also shoulder, upper arm, elbow, forearm, wrist, hand/fingers, hip/groin, thigh, knee, shinbone, ankle, and foot/toes with the response categories being right, left or both).
Pain frequency | Baseline - at time of inclusion
  Responses are presented on a 5-point Likert scale: daily, weekly, several times per week, monthly, rarely
Pain intensity: numeric pain rating scale | Baseline - at time of inclusion
  Participants are asked about worst pain during the previous week in relation to their primary pain site. Pain intensity is assessed with a 0 to 10 point numeric pain rating scale (0=no pain; 10= worst possible pain)
Pain interference | Baseline - at time of inclusion
  Participants are asked if their pain interference with their participation in E-sport (yes/no).
Eye fatigue | Baseline - at time of inclusion
  Participants are asked if they experience eye fatigue related to E-sport (yes/no).
Training load (structured E-sport) | Baseline - at time of inclusion
  Participants are asked about the number of hours they spend on structured E-sport where there is a coach present.
Training load (unstructured E-sport) | Baseline - at time of inclusion
  Participants are asked about the number of hours they spend on unstructured E-sport without a coach present.
Physical activity levels | Baseline - at time of inclusion
  International Physical Activity Questionnaire (IPAQ) short form (7 item questionnaire).
  This questionnaire assess the number of days per week spent on vigorous and moderate physical activity, walking and sitting. The questionnaire also assess the amount of time per day (hours/minutes) spent on these activities.
Hours of sleep | Baseline - at time of inclusion
  Participants are asked about how many hours they sleep on average during a night.
Trouble falling a sleep | Baseline - at time of inclusion
  Participants are asked if they have trouble falling a sleep at night (Not at all, some nights, most nights, don't know)
Waking up several times at night | Baseline - at time of inclusion
  Participants are asked if they wake up several times at night (Not at all, some nights, most nights, don't know)
Trouble sleeping through the night | Baseline - at time of inclusion
  Participants are asked if they have trouble sleeping all through the night (Not at all, some nights, most nights, don't know)
Tiered in the morning. | Baseline - at time of inclusion
  Participants are asked if they feel tiered in the morning (Not at all, some mornings, most mornings, don't know)

OTHER OUTCOMES:
Use of pain medicine | Baseline - at time of inclusion
  Participants are asked if they use pain medicine (yes/no)
Use of pain medicine - type | Baseline - at time of inclusion
  Participants are asked which type of pain medicine they use
Use of pain medicine - frequency | Baseline - at time of inclusion
  Participants are asked how frequent they use pain medicine (Several times per day, one time per day, one time per week, one time per month, rarely, don't know)
Reason for using pain medicine | Baseline - at time of inclusion
  Self-reported reason for using pain medicine
Health-care utilization | Baseline - at time of inclusion
  Participants are asked if they have sought treatment for pain from a healthcare professional during the past 3 month.

CONTACTS AND LOCATIONS:
Locations (1):
- E-Sport clubs and/or team based in the community, at an educational institution or in a private organization i Denmark, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnston R, Cahalan R, O'Keeffe M, O'Sullivan K, Comyns T. The associations between training load and baseline characteristics on musculoskeletal injury and pain in endurance sport populations: A systematic review. J Sci Med Sport. 2018 Sep;21(9):910-918. doi: 10.1016/j.jsams.2018.03.001. Epub 2018 Mar 14. PMID 29559317
- [Background] Gabbett TJ. The training-injury prevention paradox: should athletes be training smarter and harder? Br J Sports Med. 2016 Mar;50(5):273-80. doi: 10.1136/bjsports-2015-095788. Epub 2016 Jan 12. PMID 26758673
- [Background] Juho Hamari, Max Sjöblom, What is eSports and why do people watch it? Internet Res. 2017
- [Background] DiFrancisco-Donoghue J, Balentine J, Schmidt G, Zwibel H. Managing the health of the eSport athlete: an integrated health management model. BMJ Open Sport Exerc Med. 2019 Jan 10;5(1):e000467. doi: 10.1136/bmjsem-2018-000467. eCollection 2019. PMID 30792883

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT03910517/Prot_SAP_000.pdf